CLINICAL TRIAL: NCT02717130
Title: Aripiprazole, Abilify Maintena Collaborative Clinical Protocol
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated due to lack of enrollment.
Sponsor: Florida Atlantic University (Other)
Collaborators: Washington University School of Medicine (Other); University of Missouri-Columbia (Other); University of Missouri, Kansas City (Other); Burrell Behavioral Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 031-104-0014
Record Dates: First submitted 2016-03-04; First posted 2016-03-23 (Estimated); Results first posted 2020-04-13 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aripiprazole (Abilify Maintena) (Experimental): Aripiprazole once monthly (300-400 mg for entire study duration) plus 14 days oral antipsychotic medication (first injection only) (dosage according to package inserts). After the 14 day oral lead-in, after the first injection of aripiprazole once monthly, only oral aripiprazole will be allowed as a rescue medication.
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole

SUMMARY:
An Open-label, Multi-center, Longitudinal, Within-subject Comparison Study to Evaluate the Effects of Aripiprazole Once Monthly in Subjects with Schizophrenia on 30-, 90-, and 180- day Re-hospitalization Rates Following Hospital Discharge Compared with Retrospective Re-hospitalization Rates while on Oral Antipsychotic Medication.

DETAILED DESCRIPTION:
This is an open-label, multi-center, longitudinal, within-subject comparison study of the effects of aripiprazole once monthly on 30-, 90-, and 180-day psychiatric re-hospitalization rates following hospital discharge in subjects with schizophrenia compared with prior psychiatric hospitalization rates while on oral antipsychotics.

Prospective subjects will undergo screening for eligibility for entry into the study while hospitalized for symptoms due to schizophrenia.

Prospective subjects will be hospitalized for the necessary length of time as determined by the assigned treatment provider as clinically indicated, per the current standard of care. To be eligible, the anticipated duration of hospitalization should be long enough to accommodate the screening procedures, the 3-day Oral Tolerability Phase (if applicable), and initiation of treatment with aripiprazole once monthly.

During the Screening Period, subjects can be treated with any oral antipsychotic medication of the clinician's choice, with the exception of clozapine and olanzapine. However, oral olanzapine is permitted during the Screening Period only for subjects who are eligible for Phase A. Following the Screening Period, subjects who have no history of aripiprazole use will be entered into Phase A, the Oral Tolerability Phase. Subjects from Phase A that demonstrate tolerability to aripiprazole will then be entered into Phase B (i.e., the Treatment Phase). Subjects who already have a history of tolerating at least three consecutive oral doses of aripiprazole will be entered directly into Phase B. All eligible subjects will eventually enter Phase B.

Subjects who meet the inclusion and exclusion criteria and have no history of oral aripiprazole use will enter Phase A after the Screening Period while still hospitalized. Subjects in Phase A will be administered oral aripiprazole, as indicated in the product labeling, to determine tolerability. Dosage will be based on symptoms and the judgment of the investigator. The dose of oral aripiprazole may be titrated as needed. Prior antipsychotic medications will be tapered off and discontinued during the Screening Period and Phase A as clinically appropriate.

During Phase A, tolerability to oral aripiprazole will be evaluated daily for a minimum of 3 days using safety and tolerability measures (i.e., AIMS, BARS, and SAS) in conjunction with clinical judgment. If the subject shows tolerability to the oral aripiprazole, the Phase B baseline/Day 1 should occur with the first aripiprazole once monthly injection given immediately after the Phase B baseline/Day1 assessments. If a subject is unable to tolerate oral aripiprazole during the tolerability assessment in Phase A, he or she will be withdrawn from the study.

During Phase B, the subject will receive the first aripiprazole once monthly intramuscular (IM) injection, in conjunction with the first of 14 doses of concomitant oral aripiprazole, as indicated in the product labeling, after the baseline data are collected.

All subjects must attend scheduled visits at the Baseline Visit and Weeks 2, 4, 8, 12, 16, 20, and 24, totaling 180 days. Aripiprazole once monthly injections will occur at the Baseline Visit and every 28 ( -2, +5) days at Weeks 4, 8, 12, 16, 20, and 24, totaling seven injections. After the initial injection of 400 mg, the monthly dosage can be decreased to 300 mg, based on the clinical judgment of the investigator. All aripiprazole once monthly injections will be administered based on the investigator's judgment and the prescribing information.

For subjects who are psychiatrically stabilized and discharged prior to the completion of the required 14-day course of oral aripiprazole, a pre-discharge assignment will be given to a community support worker (CSW). The CSW will maintain regular contact with the subject until the first outpatient visit in Phase B (Week 2), when oral aripiprazole will be discontinued. Regular contact is defined as no less than weekly, but can be more frequent depending on the clinical judgment of the CSW and outpatient treatment team. Following the Week 2 Visit, subjects will have contact with their assigned CSW based on routine clinical care. Contact with the CSW can be in person or by telephone, as clinically appropriate.

Note: All long-acting antipsychotics are excluded from use during the study; however, aripiprazole once monthly is allowed

ELIGIBILITY:
Inclusion Criteria:

* Are able to provide written informed consent.
* Are male and female subjects 18 to 65 years of age, inclusive, at time of informed consent
* Have a current diagnosis of schizophrenia as defined by DSM-5 criteria and a history of the illness for at least 6 months prior to screening from a reliable source (e.g., subject, family member, friend, caregiver, healthcare provider, or medical records)
* Present at one of the selected inpatient units with acute psychotic symptoms for hospitalization at study entry
* Have a clinically indicated need for a change in current antipsychotic therapy
* Are on Medicaid with searchable claims data
* Have at least one inpatient psychiatric hospitalization or psychiatric ED visit within the 6 months prior to screening
* Have been previously prescribed oral antipsychotic treatment for the 6 consecutive months prior to screening
* Have a history of response to antipsychotic treatment, with no history of clozapine treatment
* Are able to understand the nature of the study and follow protocol requirements, including the prescribed dosage regimens, tablet ingestion, aripiprazole once monthly injection, and discontinuation of prohibited concomitant medications
* Are able to read and understand the written word in order to complete subject-reported outcomes measures
* Are willing to accept a monthly injection
* Are male and female subjects who are surgically sterile (i.e., have undergone orchiectomy or hysterectomy, respectively); female subjects who have been postmenopausal for at least 12 consecutive months; or male and female subjects who agree to use an approved form of birth control during study participation

Exclusion Criteria:

* Has a current DSM-5 diagnosis other than schizophrenia, including schizophreniform disorder, schizoaffective disorder, major depressive disorder, bipolar disorder, delirium, dementia, amnestic or other cognitive disorders. Also excluded are subjects with borderline, paranoid, histrionic, schizotypal, schizoid, or antisocial personality disorder.
* Prisoners or subjects who are involuntarily incarcerated, or have been incarcerated in the past 7 months for any reason
* Require potent cytochrome P450 (CYP)2D or CYP3A4 inhibitors or CYP3A4 inducers
* Are allergic, intolerant, or unresponsive to prior treatment with aripiprazole or other quinolinones or has a history of hypersensitivity to antipsychotic agents
* Have received electroconvulsive therapy within the 6 months prior to screening
* Have a history of neuroleptic malignant syndrome or clinically significant tardive dyskinesia as assessed by the investigator
* Have current diagnosis of diabetes or known fasting triglyceride levels consistent with risk for pancreatitis
* Meets DSM-5 criteria for current substance use disorder within 3 months prior to screening
* Received treatment with long-acting injectable antipsychotics (e.g., haloperidol decanoate, fluphenazine decanoate, risperidone long-acting injection [Risperdal Consta®], paliperidone palmitate extended-release injectable suspension [Invega® Sustenna®], olanzapine for extended-release injectable suspension [Zyprexa® Relprevv™]), in which the last dose was within 7 months prior to screening
* Have a significant risk of committing suicide based on history, routine psychiatric status examination, investigator's judgment, or who have an answer of "yes" on Question 4 or Question 5 within the last 30 days on the baseline version of the C-SSRS
* Have a history or evidence of a medical condition that would expose them to an undue risk of a significant AE or interfere with assessments of safety or efficacy during the course of the study, including but not limited to hepatic, renal, respiratory, cardiovascular, endocrine, neurologic, hematologic, or immunologic disease as determined by the clinical judgment of the investigator
* Have results from one or more of the following laboratory test, vital sign, and ECG tests at screening that are exclusionary (laboratory testing and ECGs will be performed locally): Platelets ≤ 75,000/mm3; Hemoglobin ≤ 9 g/dL; Fasting blood glucose > 126 mg/dL or HbA1c > 7.0%; Fasting triglyceride > 500 mg/dL; Neutrophils, absolute ≤ 1000/mm3; Aspartate transaminase (AST) > 3x ULN; Alanine transaminase (ALT) > 3x ULN; Creatinine ≥ 2 mg/dL; Diastolic blood pressure > 105 mmHg; QTc > 475 msec on either the QTcB (Bazett) or QTcF (Fridericia) corrections on ECG, confirmed by a second tracing; Any other abnormal laboratory tests, vital sign results, or ECG findings that, in the judgment of the investigator, are medically significant and would affect the safety of the subject or the interpretation of the study results. Abnormal results for laboratory parameters or vital signs should be repeated to ensure reproducibility of the abnormality before excluding a subject based on the criteria noted above.
* Have been previously enrolled in an aripiprazole once monthly clinical study
* Have participated in any clinical study with an investigational agent within the past 30 days
* Are pregnant or lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-06-08 (Actual); Primary Completion 2017-05-25 (Actual); Study Completion 2017-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Newcomer, MD, Principal Investigator — Florida Atlantic University; Ginger Nicol, MD, Principal Investigator — Washington University School of Medicine
Locations (4):
- United States (4):
  - University of Missouri, Columbia, Missouri
  - University of Missouri, Kansas City, Missouri
  - Burrell Behavioral Health, Springfield, Missouri
  - Washington University, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Covell NH, Jackson CT, Evans AC, Essock SM. Antipsychotic prescribing practices in Connecticut's public mental health system: rates of changing medications and prescribing styles. Schizophr Bull. 2002;28(1):17-29. doi: 10.1093/oxfordjournals.schbul.a006920. PMID 12047017
- [Background] Jablensky A, McGrath J, Herrman H, Castle D, Gureje O, Evans M, Carr V, Morgan V, Korten A, Harvey C. Psychotic disorders in urban areas: an overview of the Study on Low Prevalence Disorders. Aust N Z J Psychiatry. 2000 Apr;34(2):221-36. doi: 10.1080/j.1440-1614.2000.00728.x. PMID 10789527
- [Background] Barnes TR, Shingleton-Smith A, Paton C. Antipsychotic long-acting injections: prescribing practice in the UK. Br J Psychiatry Suppl. 2009 Nov;52:S37-42. doi: 10.1192/bjp.195.52.s37. PMID 19880915
- [Background] Barnes TR, Paton C, Hancock E, Cavanagh MR, Taylor D, Lelliott P; UK Prescribing Observatory for Mental Health. Screening for the metabolic syndrome in community psychiatric patients prescribed antipsychotics: a quality improvement programme. Acta Psychiatr Scand. 2008 Jul;118(1):26-33. doi: 10.1111/j.1600-0447.2008.01203.x. PMID 18582345
- [Background] Coldham EL, Addington J, Addington D. Medication adherence of individuals with a first episode of psychosis. Acta Psychiatr Scand. 2002 Oct;106(4):286-90. doi: 10.1034/j.1600-0447.2002.02437.x. PMID 12225495
- [Background] Verdoux H, Lengronne J, Liraud F, Gonzales B, Assens F, Abalan F, van Os J. Medication adherence in psychosis: predictors and impact on outcome. A 2-year follow-up of first-admitted subjects. Acta Psychiatr Scand. 2000 Sep;102(3):203-10. doi: 10.1034/j.1600-0447.2000.102003203.x. PMID 11008856
- [Background] Leucht S, Heres S. Epidemiology, clinical consequences, and psychosocial treatment of nonadherence in schizophrenia. J Clin Psychiatry. 2006;67 Suppl 5:3-8. PMID 16822090
- [Background] Thornicroft G, Farrelly S, Szmukler G, Birchwood M, Waheed W, Flach C, Barrett B, Byford S, Henderson C, Sutherby K, Lester H, Rose D, Dunn G, Leese M, Marshall M. Clinical outcomes of Joint Crisis Plans to reduce compulsory treatment for people with psychosis: a randomised controlled trial. Lancet. 2013 May 11;381(9878):1634-41. doi: 10.1016/S0140-6736(13)60105-1. Epub 2013 Mar 26. PMID 23537606
- [Background] Burns T, Rugkasa J, Molodynski A, Dawson J, Yeeles K, Vazquez-Montes M, Voysey M, Sinclair J, Priebe S. Community treatment orders for patients with psychosis (OCTET): a randomised controlled trial. Lancet. 2013 May 11;381(9878):1627-33. doi: 10.1016/S0140-6736(13)60107-5. Epub 2013 Mar 26. PMID 23537605
- [Background] Gaebel W, Schreiner A, Bergmans P, de Arce R, Rouillon F, Cordes J, Eriksson L, Smeraldi E. Relapse prevention in schizophrenia and schizoaffective disorder with risperidone long-acting injectable vs quetiapine: results of a long-term, open-label, randomized clinical trial. Neuropsychopharmacology. 2010 Nov;35(12):2367-77. doi: 10.1038/npp.2010.111. Epub 2010 Aug 4. PMID 20686456
- [Background] Olivares JM, Rodriguez-Martinez A, Buron JA, Alonso-Escolano D, Rodriguez-Morales A; e-STAR Study Group. Cost-effectiveness analysis of switching antipsychotic medication to long-acting injectable risperidone in patients with schizophrenia : a 12- and 24-month follow-up from the e-STAR database in Spain. Appl Health Econ Health Policy. 2008;6(1):41-53. doi: 10.2165/00148365-200806010-00004. PMID 18774869
- [Background] Kane JM, Carson WH, Saha AR, McQuade RD, Ingenito GG, Zimbroff DL, Ali MW. Efficacy and safety of aripiprazole and haloperidol versus placebo in patients with schizophrenia and schizoaffective disorder. J Clin Psychiatry. 2002 Sep;63(9):763-71. doi: 10.4088/jcp.v63n0903. PMID 12363115
- [Background] Potkin SG, Saha AR, Kujawa MJ, Carson WH, Ali M, Stock E, Stringfellow J, Ingenito G, Marder SR. Aripiprazole, an antipsychotic with a novel mechanism of action, and risperidone vs placebo in patients with schizophrenia and schizoaffective disorder. Arch Gen Psychiatry. 2003 Jul;60(7):681-90. doi: 10.1001/archpsyc.60.7.681. PMID 12860772
- [Background] Kasper S, Lerman MN, McQuade RD, Saha A, Carson WH, Ali M, Archibald D, Ingenito G, Marcus R, Pigott T. Efficacy and safety of aripiprazole vs. haloperidol for long-term maintenance treatment following acute relapse of schizophrenia. Int J Neuropsychopharmacol. 2003 Dec;6(4):325-37. doi: 10.1017/S1461145703003651. PMID 14609439
- [Background] Kerwin R, Millet B, Herman E, Banki CM, Lublin H, Pans M, Hanssens L, L'Italien G, McQuade RD, Beuzen JN. A multicentre, randomized, naturalistic, open-label study between aripiprazole and standard of care in the management of community-treated schizophrenic patients Schizophrenia Trial of Aripiprazole: (STAR) study. Eur Psychiatry. 2007 Oct;22(7):433-43. doi: 10.1016/j.eurpsy.2007.03.002. Epub 2007 Jun 7. PMID 17555947
- [Background] Tandon R, Devellis RF, Han J, Li H, Frangou S, Dursun S, Beuzen JN, Carson W, Corey-Lisle PK, Falissard B, Jody DN, Kujawa MJ, L'italien G, Marcus RN, McQuade RD, Ray S, Van Peborgh P; IAQ Validation Study Group. Validation of the Investigator's Assessment Questionnaire, a new clinical tool for relative assessment of response to antipsychotics in patients with schizophrenia and schizoaffective disorder. Psychiatry Res. 2005 Sep 15;136(2-3):211-21. doi: 10.1016/j.psychres.2005.05.006. PMID 16115690
- [Background] Vieta E, Bourin M, Sanchez R, Marcus R, Stock E, McQuade R, Carson W, Abou-Gharbia N, Swanink R, Iwamoto T; Aripoprazole Study Group. Effectiveness of aripiprazole v. haloperidol in acute bipolar mania: double-blind, randomised, comparative 12-week trial. Br J Psychiatry. 2005 Sep;187:235-42. doi: 10.1192/bjp.187.3.235. PMID 16135860
- [Background] Schulte RF, Boesiger P. ProFit: two-dimensional prior-knowledge fitting of J-resolved spectra. NMR Biomed. 2006 Apr;19(2):255-63. doi: 10.1002/nbm.1026. PMID 16541464
- See also: ACO #8-Risk Standardized All Condition Readmission — http://www.cms.gov/Medicare/Medicare-Fee-for-Service-Payment/sharedsavingsprogram/Downloads/Measure-ACO-8-Readmission.pdf
- See also: Outcome Measures. Baltimore: Centers for Medicare & Medicaid Services; — http://www.cms.gov/Medicare/Quality-Initiatives-Patient-Assessment-Instruments/HospitalQualityInits/OutcomeMeasures.html
- See also: Redmissions Reduction Program — http://www.cms.gov/Medicare/Medicare-Fee-for-Service-Payment/AcuteInpatientPPS/Readmissions-Reduction-Program.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aripiprazole (Abilify Maintena)
Started | 8 (Of the nine enrolled subjects, eight received study drug.)
Completed | 1
Not Completed | 7
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1
Not completed — Physician Decision | 1
Not completed — Study Closure | 4

BASELINE CHARACTERISTICS:
Arm/Group | Aripiprazole (Abilify Maintena)
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.84 (8.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 2
  African American | 6
Region of Enrollment [Number; unit: participants]
  United States | 8
Severity of Illness [Count of Participants; unit: Participants] — The Severity scale is a 7-point scale that requires the clinician to rate the severity of the patient's psychiatric illness at the time of assessment relative to the clinician's past experience with patients who have the same diagnosis. A rating of 1 corresponds to 'normal, not at all ill' patients while a rating of 7 corresponds to 'among the most extremely ill of patients'.
  Participants
    Moderately Ill | 1
    Markedly Ill | 5
    Severely Ill | 2
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per squared meter] | 29.08 (7.88)
Height [Mean (Standard Deviation); unit: centimeters] | 167.48 (13.40)
Weight [Mean (Standard Deviation); unit: kilograms] | 80.02 (16.36)
Total Cholesterol [Mean (Standard Deviation); unit: milligrams per deciliter] | 169.75 (32.38)
Triglycerides [Mean (Standard Deviation); unit: milligrams per deciliter] | 97.63 (58.34)
High-Density Lipoproteins (HDL) Cholesterol [Mean (Standard Deviation); unit: milligrams per deciliter] | 66.25 (33.97)
Low-Density Lipoproteins (LDL) Cholesterol [Mean (Standard Deviation); unit: milligrams per deciliter] | 84.13 (28.38)
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percent] | 5.11 (0.28)

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Hospital Re-admission in a 30 Day Time Frame
Description: Psychiatric re-hospitalization were planning to be assessed using hospital admission records. Study stopped due to lack of enrollment.
Time Frame: 30 days
Population: Data was not collected. The number of participants analyzed is 0 because the study was stopped due to lack of enrollment.
Arm/Group | Aripiprazole (Abilify Maintena)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: The time period over which adverse event data were collected was 30 days.
Arm/Group | Aripiprazole (Abilify Maintena)
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 3/8
Other Adverse Events (participants affected / at risk) | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole (Abilify Maintena) (N=8)
Psychiatric hospitalization (Psychiatric disorders) | 1 (2)
Seizure (Nervous system disorders) | 1 (1)
Generalized weakness (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole (Abilify Maintena) (N=8)
Prolonged QTc Interval (Cardiac disorders) | 1 (1)
Insomnia (Nervous system disorders) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
Sialorrhea (General disorders) | 1 (1)
Injection Site Pain (General disorders) | 1 (1)
Akathisia (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-26): https://cdn.clinicaltrials.gov/large-docs/30/NCT02717130/Prot_SAP_000.pdf